CLINICAL TRIAL: NCT05312268
Title: Efficacy and Safety of Rasburicase in the Treatment of Chronic Gouty Arthritis: A Multicenter Randomized Controlled Study
Brief Title: Rasburicase Treatment in Chronic Gouty Arthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KY-097-001
Record Dates: First submitted 2022-03-16; First posted 2022-04-05 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Chronic Gout
Keywords: Chronic gouty arthritis; Rasburicase
MeSH Terms: interventions — rasburicase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): Rasburicase treatment at week 1, 4 and 8 with stable dose oral urate-lowering therapy for 24 weeks.
  Interventions: Drug: Rasburicase
- Group B (Other): Rasburicase treatment at week 12, 16 and 20 with stable dose oral urate-lowering therapy for 24 weeks.
  Interventions: Drug: Rasburicase

INTERVENTIONS:
Drug: Rasburicase — Rasburicase 1.5 mg/day for 3 consecutive days at scheduled times.

SUMMARY:
The study will establish efficacy and safety of rasburicase in chronic gouty arthritis

DETAILED DESCRIPTION:
The study hypothesis is that the proportion of patients who achieved the primary endpoint after 12 weeks of treatment with rasburicase combined with oral urate-lowering therapy is superior to 12 weeks of treatment with oral urate-lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed, able to understand and comply with the requirements of the study;
* Male and female patients 18 to 70 years of age;
* Fulfill the ACR/EULAR 2015 gout classification criteria;
* Tophi detected by physical examination;
* Serum urate>300μmol/L (5mg/dl) after one-month maximum dose of urate-lowering therapy (allopurinol 600mg/d or febuxostat 80mg/d in combination with benzbromarone 100mg/d) unless intolerable OR no reduction in size of tophi after serum urate<300μmol/L (5mg/dl) for six month;

Exclusion Criteria:

* Pregnant women, lactating women, and men or women who have recently prepared for pregnancy;
* Abnormal liver function with AST, ALT, and GGT >3 times ULN;
* Blood WBC<4.0×10^9/L, and/or hemoglobin <90g/L, and/or platelets;<100×10^9/L; or other hematologic disorders;
* eGFR<15 ml/min;
* Receive following medications: azathioprine, mercaptopurine, cyclosporine, pyrazinamide, ethambutol and sulfamethoxazole
* Psychiatric disorders, history of alcoholism, drug or other substance abuse
* Immunodeficiency diseases, uncontrolled infection, etc;
* Sericosis, glucose-6-phosphate dehydrogenase activity deficiency
* Allergy to biological agents and chronic active urticaria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Monosodium urate crystal volume change evaluated by dual energy CT | Baseline to week 12 and week 12 to week 24
  Dual energy CT at baseline, week 12 and week 24

SECONDARY OUTCOMES:
Tophus volume change evaluated by physical examination | Baseline to week 12 and week 12 to week 24
The percentage of patients who have at least one tophi disappeared | Baseline to week 12 and week 12 to week 24
The percentage of patients who had achieved serum urate concentrations less than 300 μmol/L (5mg/dl) after 3 months of rasburicase treatment | Baseline to week 12 and week 12 to week 24
Number of gout flare | Baseline to week 12 and week 12 to week 24
Change of patient global assessment | Baseline to week 12 and week 12 to week 24
  The patient global assessment is given as a single question, scored from 0-10, with higher numbers representing worse perceived disease activity or overall health.
Change of physician global assessment | Baseline to week 12 and week 12 to week 24
  The physician global assessment is given as a single question, scored from 0-10, with higher numbers representing worse perceived disease activity or overall health.
Change of Visual Analog Scale (VAS) for Pain in gout flare | Baseline to week 12 and week 12 to week 24
  Visual Analog for Pain consists of a horizontal line, usually 100mm in length. The left end of the line signifies no pain while the right end signifies the worst possible pain.
Change of global functional status | Baseline to week 12 and week 12 to week 24
  The criteria are as follows: class I = able to perform usual activities of daily living (self-care, vocational, and avocational); class II = able to perform usual self-care and vocational activities, but limited in avocational activities; class III = able to perform usual self-care activities but limited in vocational and avocational activities; class IV = limited in ability to perform usual self-care, vocational, and avocational activities.
Change of Short Form 12 health survey score | Baseline to week 12 and week 12 to week 24
Change of Tophus Impact Questionnaire (TIQ)-20 score | Baseline to week 12 and week 12 to week 24
Adverse event | Baseline to week 12 and week 12 to week 24
Severe adverse event | Baseline to week 12 and week 12 to week 24
Number of patients who have positive anti-rasburicase antibodies | Baseline to week 12 and week 12 to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Qianhua Li, M.D.&Ph.D, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (4):
- China (4):
  - Shunde Hospital of Southern Medical University, Foshan, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Panyu Central Hospital, Guangzhou, Guangdong
  - Shenshan Medical Center, Shanwei, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided